CLINICAL TRIAL: NCT02508584
Title: Personalized Immunotherapeutic for Antibiotic-resistant Infection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Duane Robert Wesemann, Associate Physician and Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001027
Record Dates: First submitted 2015-07-09; First posted 2015-07-27 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Infection; Immune Deficiency; Hypogammaglobulinemia; Septic Arthritis; Mycoplasma Hominis
MeSH Terms: conditions — Infections; Immunologic Deficiency Syndromes; Agammaglobulinemia; Arthritis, Infectious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): This is a single patient treatment IND
  Interventions: Biological: anti-mycoplasma hominis antibodies

INTERVENTIONS:
Biological: anti-mycoplasma hominis antibodies — provision of customized anti-mycoplasma hominis antibodies in the context of a treatment IND.

SUMMARY:
M. A. suffers from hypogammaglobulinemia that has been complicated by refractory Mycoplasma hominis septic arthritis. He has been receiving the antibiotic valnemulin under Emergency Investigational New Drug (eIND) 114686 following many prior treatments with standard antibiotics. M.A. has also been receiving intravenous immunoglobulin (IVIG) replacement. The antibiotic and IVIG have been helpful, but not sufficient for cure. Antibodies have been shown to be critical for defense against mycoplasma. Hyperimmune serum against mycoplasma isolated from rabbit or goat has been effective in cases of chronic erosive arthritis in the setting of immune deficiency, and in some cases resulted in cures. The investigators propose to use M. hominis isolated from M. A. to vaccinate one transgenic cow (developed by SAB Biotherapeutics), purify human antibody after vaccination, test the purified antibody in killing assays to confirm potency, and then administer the purified human IgG to M. A. after FDA compassionate use IND application and local Institutional Review Board (IRB) approval.

DETAILED DESCRIPTION:
M. A. suffers from hypogammaglobulinemia that has been complicated by refractory Mycoplasma hominis septic arthritis. He has been receiving the antibiotic valnemulin under Emergency Investigational New Drug (eIND) 114686 following many prior treatments with standard antibiotics. M.A. has also been receiving intravenous immunoglobulin (IVIG) replacement. The antibiotic and IVIG have been helpful, but not sufficient for cure.

Antibodies have been shown to be critical for defense against mycoplasma. Hyperimmune serum against mycoplasma isolated from rabbit or goat has been effective in cases of chronic erosive arthritis in the setting of immune deficiency, and in some cases resulted in cures.

SAB Biotherapeutics, Inc. (formerly Sanford Applied Biosciences, LLC) located in Sioux Falls, SD, have developed transchromosomic (Tc) cows containing human immunoglobulin (Ig) heavy (IgH) and light (IgL) chain loci in the setting of inactivated bovine IgH and Ig lambda loci. To date, SAB Biotherapeutics (SAB) has several products in development that have been tested in animal models, but to date no human trials.

Investigators propose to use M. hominis isolated from M. A. to vaccinate one transgenic cow, purify antibody after vaccination, test the purified antibody in killing assays to confirm potency, and then administer the purified human IgG to M. A. after FDA compassionate use IND application and local Institutional Review Board (IRB) approval.

M. A. is a highly educated person with full decision making capacity and is well aware of the uncertainties and risks associated with this treatment. This proposal is designed to offer this patient an alternative and perhaps curative approach to his disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult with decision making capacity afflicted with chronic mycoplasma hominis septic arthritis despite standard treatments.

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Presence or absence of mycoplasma hominis cultured from joint and wound fluid | from date of initiation of therapy up to 1 year
  see publication below
Patency of fistula as assessed by clinical exam | from date of initiation of therapy up to 1 year
  see publication below
Pain reduction as measured by pain scale and amount of pain medication required | from date of initiation of therapy up to 1 year
  see publication below

CONTACTS AND LOCATIONS:
Overall Officials: Duane R. Wesemann, MD, PhD, Principal Investigator — Brigham and Women's Hosptial
Locations (1):
- Brigham and Women's Hosptial, Boston, Massachusetts, United States

REFERENCES:
- [Result] Silver JN, Ashbaugh CD, Miles JJ, Wu H, Marecki GT, Hwang JK, Jiao JA, Abrams M, Sullivan EJ, Wesemann DR. Deployment of Transchromosomal Bovine for Personalized Antimicrobial Therapy. Clin Infect Dis. 2018 Mar 19;66(7):1116-1119. doi: 10.1093/cid/cix977. PMID 29272362